CLINICAL TRIAL: NCT03687177
Title: Visual Cue as Prevention of Pulmonary Infection Under Mechanical Ventilation
Acronym: PREVIP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 6793
Record Dates: First submitted 2018-09-25; First posted 2018-09-27 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Pulmonary Infection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): Nurses from intensive care informed on the prevention of VAP and without visual cue to estimate the angle of elevation of the head of intubated patients
  Interventions: Other: Without visual cue and nurses informed
- Experimental group (Other): Nurses from intensive care informed on the prevention of VAP with visual cue to estimate the angle of elevation of the head of intubated patients.
  Interventions: Other: With visual cue and nurses informed

INTERVENTIONS:
Other: With visual cue and nurses informed — Using visual cue or no visual cue with to estimate the angle of elevation of the head of intubated patients with prevention of nurse
  Arms: Experimental group
Other: Without visual cue and nurses informed — Not using visual cue or no visual cue with to estimate the angle of elevation of the head of intubated patients with prevention of nurse
  Arms: Control group

SUMMARY:
Nosocomial pneumonia is the third causes of nosocomial infection. In intensive care unit, their incidence is even higher, of the order of 10 to 30% in patients with invasive mechanical ventilation (IMV). One of the main mechanisms behind VAP (Ventilator-Associated Pneumonia) is the passage of germs colonizing the oropharynx to the subglottic airways. The presence of a nasogastric tube, immobilization, and strict dorsal decubitus increase the risk of colonization of the tracheobronchial tree and pneumonia in these patients. To reduce the incidence of VAP, several strategies have been developed in intensive care to try to control these different risk factors. These sets of measures, also called "bundle" systematically include the control of the elevation of the patient's head more than 30 °. Nevertheless, the strict and permanent control of the elevation of the patient's head is difficult to obtain. One of the reasons that may explain the difficulty of ensuring a correct elevation is the absence of visual cues that are easy to obtain on the beds of patients. An easily identifiable visual cue at the head of the bed would probably provide a satisfactory elevation (greater than 30 °) in patients intubated in intensive care. Our hypothesis is that the addition to the head of the patient's bed of a visible mark that is easily visible and easily interpretable by all the nurses will improve the elevation of the head of the patients in intensive care.

ELIGIBILITY:
Inclusion Criteria:

- Patient admitted to intensive care with invasive mechanical ventilation more than two days

Exclusion Criteria:

* Pregnancy
* Spinal trauma
* Brain trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2018-09-20 (Actual); Primary Completion 2019-10-22 (Estimated); Study Completion 2019-10-22 (Estimated)

PRIMARY OUTCOMES:
Measurement of the angle of elevation of the head of patients with invasive mechanical ventilation | 3 times a day

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France